CLINICAL TRIAL: NCT01441596
Title: Lux-Breast 3; Randomised Phase II Study of Afatinib Alone or in Combination With Vinorelbine Versus Investigator's Choice of Treatment in Patients With HER2 Positive Breast Cancer With Progressive Brain Metastases After Trastuzumab and/or Lapatinib Based Therapy
Brief Title: Lux-Breast 3; Afatinib Alone or in Combination With Vinorelbine in Patients With Human Epidermal Growth Factor Receptor 2 (HER2) Positive Breast Cancer Suffering From Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200.67; 2010-021415-16 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-09-26; First posted 2011-09-27 (Estimated); Results first posted 2015-02-25 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-08

CONDITIONS: Breast Neoplasms; Neoplasm Metastasis
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Vinorelbine; Afatinib

ARMS (3):
- arm A: Afatinib monotherapy (Experimental): Afatinib monotherapy: starting dose 40 mg per day, continuous treatment in a 3-weekly course. If well tolerated, the dose may be escalated to 50 mg.
  Interventions: Drug: afatinib
- arm B: Afatinib in combination with vino (Experimental): Afatinib 40 mg per day, continuous treatment, in combination with vinorelbine Vinorelbine 25 mg/mÂ² on days 1, 8, 15 in a 3-weekly course.
  Interventions: Drug: Vinorelbine; Drug: afatinib
- arm C: investigator's choice of treatmen (Active Comparator): Patients will receive, at the investigator's discretion, the most appropriate medical treatment consisting of single agent or combination regimen approved for the treatment of metastatic breast cancer, and according to patient status and local guidelines.
  Interventions: Drug: Investigator's choice of treatment

INTERVENTIONS:
Drug: Vinorelbine — Vinorelbine 25 mg/mÂ² on days 1, 8, 15 in a 3-weekly course
  Arms: arm B: Afatinib in combination with vino
Drug: Investigator's choice of treatment — Patients will receive, at the investigator's discretion, the most appropriate medical treatment consisting of single agent or combination regimen approved for the treatment of metastatic breast cancer, and according to patient status and local guidelines.
  Arms: arm C: investigator's choice of treatmen
Drug: afatinib — Afatinib monotherapy:once daily, continuous treatment in a 3-weekly course. If well tolerated, the dose may be escalated to 50 mg.
  Arms: arm B: Afatinib in combination with vino
Drug: afatinib — Afatinib monotherapy:once daily, continuous treatment in a 3-weekly course. If well tolerated, the dose may be escalated to 50 mg.
  Arms: arm A: Afatinib monotherapy

SUMMARY:
The aim of this study is to investigate the efficacy and safety of afatinib alone or in combination with vinorelbine, as treatment in patients with HER2-overexpressing metastatic breast cancer, who have progressive brain lesions after trastuzumab and/or lapatinib based therapy

ELIGIBILITY:
Inclusion criteria:

1. patients with HER2 positive breast cancer with a documented central nervous system (CNS) recurrence/progression (by imaging) during or after a HER2 inhibitor (Trastuzumab and/or Lapatinib) based therapy (no leptomeningeal carcinomatosis as the only site of CNS metastases)
2. at least one measurable and progressive lesion in the brain (=10 mm on T1-weighted, gadolinium-enhanced Magnetic Resonance Imaging). Measurable or non measurable extracranial metastases allowed.
3. previous treatment with HER2 inhibitors to be discontinued prior to first study treatment administration (at least 14 days for trastuzumab and other antibodies, at least 7 days for lapatinib).
4. previous chemotherapy and hormonal therapy (adjuvant and metastatic regimens) allowed, but chemotherapy must have been discontinued at least 14 days and hormonal therapy at least 7 days prior to first study treatment administration.
5. Patients must have recovered to baseline condition or to Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 grade = 1 from any acute CTCAE v. 3.0 grade =2 side effects of previous treatments.
6. prior surgery, whole brain radiotherapy or stereotactic radiosurgery allowed provided that there is unequivocal evidence of one or more new and/or progressive brain metastases after completion of whole brain radiotherapy or stereotactic radiosurgery.

Exclusion criteria:

1. Prior treatment with HER2- tyrosine kinase inhibitor other than lapatinib
2. Any other current malignancy or malignancy diagnosed within the past five (5) years (other than bilateral primary breast cancer, metastases to the contralateral breast, non-melanomatous skin cancer and in situ cervical cancer).
3. Significant chronic or recent acute gastrointestinal disorders with diarrhoea as a major symptom e.g. Crohn's disease, malabsorption or Common Terminology Criteria (CTC) grade =2 diarrhoea of any aetiology.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2011-10; Primary Completion 2014-02 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (40):
- United States (6):
  - 1200.67.10106 Boehringer Ingelheim Investigational Site, Bakersfield, California
  - 1200.67.10105 Boehringer Ingelheim Investigational Site, Fullerton, California
  - 1200.67.10001 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1200.67.10108 Boehringer Ingelheim Investigational Site, Santa Barbara, California
  - 1200.67.10003 Boehringer Ingelheim Investigational Site, Lake Success, New York
  - 1200.67.10004 Boehringer Ingelheim Investigational Site, Columbus, Ohio
- Canada (3):
  - 1200.67.11004 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1200.67.11003 Boehringer Ingelheim Investigational Site, Greenfield Park, Quebec
  - 1200.67.11002 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- Finland (3):
  - 1200.67.35801 Boehringer Ingelheim Investigational Site, Helsinki
  - 1200.67.35802 Boehringer Ingelheim Investigational Site, Tampere
  - 1200.67.35803 Boehringer Ingelheim Investigational Site, Turku
- France (10):
  - 1200.67.33009 Boehringer Ingelheim Investigational Site, Caen
  - 1200.67.33010 Boehringer Ingelheim Investigational Site, Clermont-Ferrand
  - 1200.67.33008 Boehringer Ingelheim Investigational Site, Lille
  - 1200.67.33001 Boehringer Ingelheim Investigational Site, Lyon
  - 1200.67.33004 Boehringer Ingelheim Investigational Site, Marseille
  - 1200.67.33011 Boehringer Ingelheim Investigational Site, Nice
  - 1200.67.33002 Boehringer Ingelheim Investigational Site, Paris
  - 1200.67.33003 Boehringer Ingelheim Investigational Site, Paris
  - 1200.67.33012 Boehringer Ingelheim Investigational Site, Saint-Cloud
  - 1200.67.33005 Boehringer Ingelheim Investigational Site, Saint-Herblain
- Germany (7):
  - 1200.67.49002 Boehringer Ingelheim Investigational Site, Erlangen
  - 1200.67.49008 Boehringer Ingelheim Investigational Site, Essen
  - 1200.67.49005 Boehringer Ingelheim Investigational Site, Hanover
  - 1200.67.49006 Boehringer Ingelheim Investigational Site, Heidelberg
  - 1200.67.49007 Boehringer Ingelheim Investigational Site, MÃ¼nchen
  - 1200.67.49003 Boehringer Ingelheim Investigational Site, Oldenburg
  - 1200.67.49004 Boehringer Ingelheim Investigational Site, TÃ¼bingen
- Italy (2):
  - 1200.67.39001 Boehringer Ingelheim Investigational Site, Modena
  - 1200.67.39002 Boehringer Ingelheim Investigational Site, Reggio Emilia
- South Korea (4):
  - 1200.67.82001 Boehringer Ingelheim Investigational Site, Goyang
  - 1200.67.82002 Boehringer Ingelheim Investigational Site, Seoul
  - 1200.67.82003 Boehringer Ingelheim Investigational Site, Seoul
  - 1200.67.82004 Boehringer Ingelheim Investigational Site, Seoul
- Spain (5):
  - 1200.67.34002 Boehringer Ingelheim Investigational Site, Barcelona
  - 1200.67.34006 Boehringer Ingelheim Investigational Site, CÃ³rdoba
  - 1200.67.34005 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat
  - 1200.67.34003 Boehringer Ingelheim Investigational Site, Madrid
  - 1200.67.34004 Boehringer Ingelheim Investigational Site, Valencia

REFERENCES:
- [Derived] Cortes J, Dieras V, Ro J, Barriere J, Bachelot T, Hurvitz S, Le Rhun E, Espie M, Kim SB, Schneeweiss A, Sohn JH, Nabholtz JM, Kellokumpu-Lehtinen PL, Taguchi J, Piacentini F, Ciruelos E, Bono P, Ould-Kaci M, Roux F, Joensuu H. Afatinib alone or afatinib plus vinorelbine versus investigator's choice of treatment for HER2-positive breast cancer with progressive brain metastases after trastuzumab, lapatinib, or both (LUX-Breast 3): a randomised, open-label, multicentre, phase 2 trial. Lancet Oncol. 2015 Dec;16(16):1700-10. doi: 10.1016/S1470-2045(15)00373-3. Epub 2015 Nov 17. PMID 26596672

RESULTS

PARTICIPANT FLOW:
Groups:
- Afatinib Mono: Afatinib monotherapy administered orally: starting dose 40 mg per day, continuous treatment in a 3-weekly course. If well tolerated, the dose may be escalated to 50 mg.
- Afatinib+Vino: Afatinib 40 mg per day administered orally, continuous treatment, in combination with weekly Vinorelbine 25 mg/m² administered intravenously on days 1, 8, 15 in a 3-weekly course.
- Investigator's Choice: Patients will receive, at the investigator's discretion, the most appropriate medical treatment consisting of single agent or combination regimen approved for the treatment of metastatic breast cancer, and according to patient status and local guidelines.
Period: Overall Study
Arm/Group | Afatinib Mono | Afatinib+Vino | Investigator's Choice
Started | 40 | 38 | 43
Completed | 36 | 35 | 39
Not Completed | 4 | 3 | 4
Not completed — Other reason not defined below | 0 | 2 | 1
Not completed — Withdrawal by Subject | 4 | 0 | 2
Not completed — Not treated | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomised Set (RS): includes all randomised patients, whether treated or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib Mono | Afatinib+Vino | Investigator's Choice | Total
Number analyzed (Participants) | 40 | 38 | 43 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (10.3) | 51.2 (10.6) | 52.6 (10.3) | 51.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 38 | 43 | 121
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Patient Benefit Rate at 12 Weeks
Description: Percentage of patients with patient benefit at week 12. Patient benefit was defined by the absence of central nervous system (CNS) disease progression according to Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1 in addition to no tumour-related worsening of the neurological signs and symptoms (NSS), no tumour-related increase in corticosteroid dosage and no progression of extra CNS disease according to RECIST 1.1
Time Frame: 12 weeks from randomisation
Population: Randomised Set (RS): includes all randomised patients, whether treated or not.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Afatinib Mono | Afatinib+Vino | Investigator's Choice
Number analyzed (Participants) | 40 | 38 | 43
percentage of participants | 30.0 [16.6 to 46.5] | 34.2 [19.6 to 51.4] | 41.9 [27.0 to 57.9]

2. Secondary Outcome: Progression-Free Survival
Description: Progression-Free Survival is defined as the time from the date of randomisation to the date of disease progression or death whichever came first.
  Disease progression was defined as either disease progression in CNS lesions (including worsening in NSS and use of corticosteroid) or disease progression in extra-CNS lesions according to RECIST 1.1.
Time Frame: From first drug administration until 28 days after end of treatment, up to 805 days
Population: RS including only patients who experienced disease progression or death
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Afatinib Mono | Afatinib+Vino | Investigator's Choice
Number analyzed (Participants) | 40 | 38 | 43
weeks | 11.9 [6.1 to 20.9] | 12.3 [6.3 to 23.3] | 18.4 [8.3 to 30.7]

3. Secondary Outcome: Overall Survival
Description: Overall Survival is defined as time from randomisation to the date of death from any cause.
Time Frame: From first drug administration until 28 days after end of treatment, up to 805 days
Population: RS including only patients who died
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Afatinib Mono | Afatinib+Vino | Investigator's Choice
Number analyzed (Participants) | 40 | 38 | 43
weeks | 57.7 [34.1 to 81.3] | 37.3 [21.0 to 66.7] | 52.1 [29.1 to 122.6]

ADVERSE EVENTS:
Time Frame: From first drug administration until 28 days after end of treatment, up to 805 days
Arm/Group | Afatinib Mono | Afatinib+Vino | Investigator's Choice
Serious Adverse Events (participants affected / at risk) | 18/40 | 24/37 | 22/42
Other Adverse Events (participants affected / at risk) | 39/40 | 37/37 | 40/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib Mono (N=40) | Afatinib+Vino (N=37) | Investigator's Choice (N=42)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 1
Progressive cerebellar degeneration (Congenital, familial and genetic disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 5 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2 | 1
Asthenia (General disorders) | 0 | 2 | 1
Chest discomfort (General disorders) | 0 | 1 | 0
Concomitant disease progression (General disorders) | 0 | 1 | 1
Death (General disorders) | 0 | 0 | 2
General physical health deterioration (General disorders) | 4 | 6 | 1
Generalised oedema (General disorders) | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 0
Device related infection (Infections and infestations) | 0 | 2 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 3 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1
Septic shock (Infections and infestations) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0
Brain herniation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
CSF protein increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 2 | 3 | 3
Dizziness (Nervous system disorders) | 1 | 2 | 1
Epilepsy (Nervous system disorders) | 2 | 1 | 0
Headache (Nervous system disorders) | 0 | 3 | 2
Hemiparesis (Nervous system disorders) | 0 | 1 | 0
Hemiplegia (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Motor dysfunction (Nervous system disorders) | 0 | 0 | 1
Motor neurone disease (Nervous system disorders) | 1 | 0 | 0
Neurological symptom (Nervous system disorders) | 0 | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 2
Mood altered (Psychiatric disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib Mono (N=40) | Afatinib+Vino (N=37) | Investigator's Choice (N=42)
Anaemia (Blood and lymphatic system disorders) | 1 | 12 | 6
Leukopenia (Blood and lymphatic system disorders) | 0 | 3 | 5
Lymphopenia (Blood and lymphatic system disorders) | 1 | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 23 | 11
Vertigo (Ear and labyrinth disorders) | 1 | 6 | 9
Diplopia (Eye disorders) | 0 | 0 | 5
Dry eye (Eye disorders) | 1 | 4 | 3
Vision blurred (Eye disorders) | 3 | 4 | 4
Visual impairment (Eye disorders) | 3 | 5 | 5
Abdominal distension (Gastrointestinal disorders) | 2 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 6 | 7
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 1
Constipation (Gastrointestinal disorders) | 8 | 10 | 14
Diarrhoea (Gastrointestinal disorders) | 36 | 31 | 16
Dry mouth (Gastrointestinal disorders) | 2 | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 2 | 2
Gastritis (Gastrointestinal disorders) | 0 | 3 | 0
Haemorrhoids (Gastrointestinal disorders) | 4 | 1 | 1
Nausea (Gastrointestinal disorders) | 10 | 13 | 15
Stomatitis (Gastrointestinal disorders) | 5 | 13 | 6
Vomiting (Gastrointestinal disorders) | 7 | 9 | 11
Asthenia (General disorders) | 11 | 9 | 14
Fatigue (General disorders) | 8 | 11 | 3
Gait disturbance (General disorders) | 2 | 3 | 1
Malaise (General disorders) | 0 | 2 | 0
Mucosal inflammation (General disorders) | 8 | 11 | 6
Oedema peripheral (General disorders) | 4 | 2 | 5
Pain (General disorders) | 1 | 3 | 2
Pyrexia (General disorders) | 0 | 2 | 3
Xerosis (General disorders) | 0 | 2 | 0
Bronchitis (Infections and infestations) | 3 | 1 | 1
Conjunctivitis (Infections and infestations) | 4 | 2 | 0
Cystitis (Infections and infestations) | 0 | 3 | 2
Paronychia (Infections and infestations) | 5 | 6 | 1
Rhinitis (Infections and infestations) | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 8 | 6
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 3
Alanine aminotransferase increased (Investigations) | 1 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 0
Weight decreased (Investigations) | 2 | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 9 | 9 | 10
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 7 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 6 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2
Aphasia (Nervous system disorders) | 1 | 3 | 3
Ataxia (Nervous system disorders) | 2 | 3 | 4
Balance disorder (Nervous system disorders) | 1 | 2 | 2
Brain oedema (Nervous system disorders) | 0 | 2 | 0
Dizziness (Nervous system disorders) | 8 | 9 | 12
Dysarthria (Nervous system disorders) | 1 | 3 | 1
Headache (Nervous system disorders) | 11 | 11 | 16
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 4
Neurotoxicity (Nervous system disorders) | 3 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2 | 3
Somnolence (Nervous system disorders) | 3 | 3 | 1
Tremor (Nervous system disorders) | 0 | 1 | 3
Anxiety (Psychiatric disorders) | 2 | 2 | 2
Depression (Psychiatric disorders) | 1 | 2 | 1
Insomnia (Psychiatric disorders) | 6 | 5 | 4
Dysuria (Renal and urinary disorders) | 1 | 3 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3 | 8
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 8 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 5 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 2 | 2
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 | 0 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 15 | 20 | 4
Skin lesion (Skin and subcutaneous tissue disorders) | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.